CLINICAL TRIAL: NCT07011576
Title: A Phase II Study Investigating Fruquintinib Plus FOLFIRI as Second-Line Treatment for Participants With Metastatic Colorectal Cancer (mCRC)
Brief Title: A Study of Fruquintinib Plus FOLFIRI as Second-Line Treatment for Participants With Metastatic Colorectal Cancer (mCRC)
Acronym: FRUITFUL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Takeda Development Center Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GI 387
Record Dates: First submitted 2025-06-05; First posted 2025-06-09 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Colon Cancer; Rectal Cancer; Colorectal Cancer; Colorectal Cancer (CRC)
Keywords: Colorectal cancer; Colon Cancer; Rectal cancer; Metastatic colorectal cancer; mCRC; VEGFR inhibitor; Fruquintinib; FOLFIRI; Second line; 2L mCRC
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms; Colorectal Neoplasms | interventions — HMPL-013; Irinotecan; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Fruquinitinib + FOLFIRI (Experimental): Participants will receive an assigned dose level of fruquintinib in combination with FOLFIRI. Cycles will be 28 days, where participants will take fruquinitinib orally on Days 1 through 21 in combination with FOLFIRI intravenous infusion (IV) every 2 weeks. Up to 60 participants will be enrolled.
  Interventions: Drug: fruquintinib; Drug: FOLFIRI (Irinotecan, 5-Fluorouracil, and Leucovorin)

INTERVENTIONS:
Drug: fruquintinib — Participants will receive oral fruquintinib, with or without food, for the first 21 days of each 28-day cycle.
  Other Names: Fruzaqla
Drug: FOLFIRI (Irinotecan, 5-Fluorouracil, and Leucovorin) — Participants will receive FOLFIRI once every 2 weeks on day 1 of every 28-day cycle (twice in each cycle). The FOLFIRI regimen consists of irinotecan given 180 mg/m2 intravenous infusion (IV), leucovorin 400 mg/m2 (or 200 mg/m2 levoleucovorin) IV, followed by 5-fluorouracil (5-FU) 400 mg/m2 bolus injection and 5-FU continuous IV infusion of 2400 mg/m2 over 46 to 48 hours.

SUMMARY:
This is an open-label multicenter, single-arm Phase II study of Fruquintinib in combination with FOLFIRI (leucovorin calcium (folinic acid), fluorouracil, and irinotecan) in participants with metastatic colorectal cancer (mCRC). The main goals of this study are to:

* Evaluate the efficacy of the combination of fruquintinib + FOLFIRI in the 2nd-line mCRC setting
* Evaluate the safety of the combination of fruquintinib + FOLFIRI

DETAILED DESCRIPTION:
Fruquintinib is an FDA approved cancer medication that works by targeting proteins called vascular endothelial growth factor receptors (VEGFRs). VEGFRs are important in the creation of new blood vessels. As a highly-selective and potent VEGFR inhibitor, fruquintinib helps block new blood vessels that would provide nutrients and oxygen to cancerous tumors from forming. It is a small molecule anti-tumor drug with a novel chemical structure that belongs to the quinazoline class.

This study is an open-label Phase II study designed to evaluate the efficacy and safety of fruquintinib + FOLFIRI in 2nd-line setting mCRC participants who have been previously treated with FOLFOX (folinic acid, fluorouracil, and oxaliplatin) and Bevacizumab-based first-line therapy. Up to 60 participants will receive concurrent fruquintinib and FOLFIRI according to standard guidelines of treatment of mCRC.

ELIGIBILITY:
Key Inclusion Criteria:

* Confirmed mCRC ; histologically documented adenocarcinoma of the colon or rectum with at least one measurable lesion according to RECIST v1.
* Genetic aberrations are allowed, except for microsatellite instability high (MSI-H) and BRAF V600
* Participants must have received FOLFOX (folinic acid, fluorouracil, and oxaliplatin) and Bevacizumab- based first-line therapy for mCRC
* At least 18 years-of-age at the time of signature of the Informed Consent Form (ICF)
* Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 to 2

Key Exclusion Criteria:

* Current treatment with other anticancer treatments within 21 days of the first dose of study treatment
* Major surgery within 4 weeks of the first planned dose of study treatment
* More than one treatment received for mCRC prior to signing the ICFs
* Uncontrolled, symptomatic brain metastases
* Uncontrolled, symptomatic gastrointestinal disease
* Patients with uncontrolled hypertension
* Women who are pregnant, nursing, or plan to become pregnant while in the study and for at least 6 months after the last administration of study chemotherapy
* Men who plan to father a child while in the study and for at least 6 months after the last administration of study chemotherapy
* Documented major electrocardiogram (ECG) abnormalities which are clinically significant.
* Symptomatic or uncontrolled brain metastases, spinal cord compression, or leptomeningeal disease requiring concurrent treatment
* Presence of other active invasive cancers other than the one treated in this study within 5 years prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-29 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) rate at 6 months | Every 2 cycles from cycle 1 day 1, until disease progression or death, up to 2 years. Each cycle is 28 days.
  Progression-Free Survival (PFS) rate at 6 months, defined as the percentage of participants at 6 months who have not experienced disease progression as defined by the RECIST Version 1.1 criteria or death on study. Participants who are alive and free from disease progression will be censored at the date of last tumor assessment.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Every 2 cycles from cycle 1 day 1, until disease progression or death, up to 2 years. Each cycle is 28 days.
  Objective Response Rate (ORR), defined as the proportion of participants with confirmed CR or PR (i.e., 2 CRs or PRs at least 4 weeks apart) according to the RECIST Version 1.1.
Duration of response (DoR) | Every 2 cycles from cycle 1 day 1, until disease progression or death, up to 2 years. Each cycle is 28 days.
  Duration of Response (DoR), defined as the duration from the first documented response to the date of first documented PD or death due to any cause. In case a participant does not experience PD or death, DoR is censored at the date of last adequate tumor assessment (defined as an assessment of CR, PR, or SD). DoR analysis will include only responders (PR or better).
Disease control response rate (DCR) | Every 2 cycles from cycle 1 day 1, until disease progression or death, up to 2 years. Each cycle is 28 days.
  Disease Control Response Rate (DCR), defined as the proportion of participants with a best overall response of CR, PR, or SD.
Number of participants with treatment emergent adverse events | Every 28 day cycle, from signed informed consent to 30 days after treatment discontinuation up to 1 year.
  Using CTCAE V5.0
Overall Survival (OS) | From cycle 1 day 1 up to 2 years
  Overall Survival (OS), defined as the time from the first day of study drug administration (Day 1) to death. Participants who are alive will be censored at the date of last known date alive. Each cycle is 28 days.

CONTACTS AND LOCATIONS:
Overall Officials: Meredith Pelster, MD, Study Chair — SCRI Oncology Partners
Locations (11):
- United States (11):
  - Rocky Mountain Cancer Center - Primary, Denver, Colorado
  - Maryland Oncology Hematology, Columbia, Maryland
  - Minnesota Oncology Hematology - Primary, Maple Grove, Minnesota
  - Oncology Associates of Oregon - Primary, Eugene, Oregon
  - Northwest Cancer Specialists - Compass, Portland, Oregon
  - SCRI Oncology Partners, Nashville, Tennessee
  - Texas Oncology - Central/South Texas, Austin, Texas
  - Texas Oncology - Gulf Coast, Beaumont, Texas
  - Texas Oncology - Northeast Texas, Tyler, Texas
  - Virginia Oncology Associates, Norfolk, Virginia
  - Blue Ridge Cancer Care (Oncology & Hematology Associates of Southwest VA), Salem, Virginia